CLINICAL TRIAL: NCT01591239
Title: Parents as Interventionists for Moderate Drug Abusing Adolescents
Brief Title: Home-Based Program to Help Parents of Drug Abusing Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: University of Minnesota (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50DA027841 (NIH); P50DA027841 (NIH)
Record Dates: First submitted 2012-04-07; First posted 2012-05-03 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Substance-Related Disorders; Drug Addiction; Substance Abuse
Keywords: Adolescent; Parent; Substance Abuse; Parent Training; Addiction; Family Intervention; Brief Intervention; Home Intervention
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-Based Intervention (Experimental): Parents will receive a 1-session training on how to deliver a 3-session intervention across a 3-week period. The intervention program begins with a 3 and a half hour training session delivered by the staff Trainer to the participating parent. At the conclusion of training, the parent will be given the intervention manual and supplemental materials. The trainer will phone the parent shortly before session 1, in between each intervention session, and after the third intervention (four phone calls total) to review the objectives and tasks associated with that week's intervention session and to help prepare for the coming session. At the final phone call between the parent and trainer (after the third week), the trainer will deliver to the parent the follow-up resources.
  Interventions: Behavioral: Home-Based Intervention
- Educational Group (Active Comparator): Parents will receive a 2-hour, education-only psychoeducational curriculum (no parent-led intervention with their teen will occur.
  Interventions: Behavioral: Educational Group

INTERVENTIONS:
Behavioral: Home-Based Intervention — Parents will be trained through a 3 1/2-hour series on providing a 3-session drug and alcohol intervention program to their adolescent. The parent-led intervention will require parents to meet with their adolescent and work together to help strengthen family cohesiveness, enhance communication, and promote healthy life choices.
  Arms: Home-Based Intervention
Behavioral: Educational Group — Printed fact sheets will be delivered to parents in a single two-hour session. These fact sheets will provide general drug-related information from the public domain (e.g., substance use trends and well-known dangers of substance involvement), and focus on communication approaches and talking points when discussing substance use with their adolescent (e.g., why adolescents use; how the media may influence attitudes about substances).
  Arms: Educational Group

SUMMARY:
This project is aimed at parents with a teenager who is already starting to use drugs. The study will test a new, innovative version of a brief intervention. This program will be home based rather than implemented by a counselor in a clinical setting. The stage I activities will involve manual development, parent training development, and a small feasibility study; Stage II involves an efficacy study. Two samples, 110 families each, will participate in the trial. Families will be assigned to either an intervention or control condition. The investigators hypothesize that the home-based intervention will be superior to the control condition. In addition, the investigators expect response to the intervention by the adolescent to be mediated by motivation, cognitions, problem solving, peer drug use, parenting skills and parent self-efficacy.

DETAILED DESCRIPTION:
Little attention has been paid to the large group of adolescents who use substances but are not, or not yet, dependent and who could successfully reduce substance use through early intervention. Brief interventions (BI) that are based in cognitive-behavioral and motivational interviewing (CB-MI) strategies provide an option for such mid-level drug abusers (e.g., DSM-IV substance abuse disorder), and extant research on them suggests this approach can be effective with youth.

Winters and colleagues have studied with controlled designs the efficacy of brief interventions for application to mild-to-moderate substance abusing adolescents. These studies have used the more traditional approach of counselor-led interventions. This program will be parent-led rather than directed by a counselor in a clinical setting.

The stage I activities will involve manual development, parent training development, and a small feasibility study; Stage II involves an efficacy trial. Two samples, 110 families each, will participate in the trial. Families will be assigned to either an intervention or control condition. Data to quantify intervention effects will be obtained by interviewing adolescents and the target parent at multiple time points (baseline and, 3-, 6- and 12-months post baseline). The investigators hypothesize that the home-based intervention will be superior to the control condition. In addition, the investigators expect response to the intervention by the adolescent to be mediated by motivation, cognitions, problem solving, peer drug use, parenting skills and parent self-efficacy. Secondary analyses will focus on additional predictors of intervention effects, and analyses of parent adherence, parent acceptance, and of training adherence.

The final product of the work will be a tested comparative intervention protocol that is shaped in an engaging and useful presentation format for use by parents.

ELIGIBILITY:
Inclusion Criteria:

1. Referral of the adolescent to the Minneapolis metro area participating sites.
2. Both the parent and teen consent to participate.

Exclusion Criteria:

1. Current developmental disorder or learning disorder.
2. current or past history of psychosis, or any psychiatric or other condition that may interfere with ongoing participation in the intervention.
3. Suicidal ideation or otherwise judged to be at risk to self or others
4. Unstable or uncontrolled medical illnesses which may interfere with participation in the study.
5. Inability to understand the study procedures or otherwise give informed assent for participation.
6. Failure by the parent to give informed consent for the adolescent.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adolescent Substance Use | Changes from Baseline at 3-, 6-, and 12- months post-baseline
  Adolescent participants will complete the Timeline Follow Back in order to assess days of drug use.
Adolescent Drug Use Consequences | Changes from Baseline at 3-, 6-, and 12- months post-baseline
  The adolescent participant will complete the Personal Consequences Scale in order to measure their drug use consequences.
DSM-IV Substance Use Diagnosis | Changes from Baseline at 3-, 6-, and 12- months post-baseline
  The Adolescent Diagnostic Interview (ADI) will be used to determine a diagnosis.

SECONDARY OUTCOMES:
Adolescent Mental Health | Baseline and 3-, 6-, and 12- months post-baseline
  Adolescent mental health will be measured in two ways. The parent participant will complete the ADI-Parent version and the adolescent participant will complete the Comprehensive Adolescent Severity Inventory (CASI).
Adolescent Treatment History | Baseline and 3-, 6-, and 12- months post-baseline
  Parent participants will provide this data when completing the ADI-Parent version.
Program Acceptability | Parent Training (average of 2 weeks post-baseline) and Post-Session 3 (average of 6 weeks after the parent training)
  The Credibility/Expectancy Questionnaire (CEQ) will be completed by parents during the training session and the Working Alliance Inventory (WAI) will be completed my the parent after he or she completes the third training session with the adolescent.
Program Satisfaction | Post-Session 3 (average of 6 weeks after the parent training)
  Parents will complete a satisfaction questionnaire after completing the third session with the adolescent participant.
Training Fidelity | Parent Training (average of 2 weeks post-baseline)
  A training fidelity checklist will be completed by an assessor following the training.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Winters, Ph.D., Principal Investigator — Treatment Research Institute and University of Minnesota
Locations (1):
- University of Minnesota Medical School, Department of Psychiatry, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Botzet AM, Dittel C, Birkeland R, Lee S, Grabowski J, Winters KC. Parents as interventionists: Addressing adolescent substance use. J Subst Abuse Treat. 2019 Apr;99:124-133. doi: 10.1016/j.jsat.2019.01.015. Epub 2019 Jan 23. PMID 30797384